CLINICAL TRIAL: NCT00063752
Title: An Open-Label, Dose-Escalation, Phase I Clinical Study to Assess the Safety of PI-0824 in Patient With Pemphigus Vulgaris Requiring Daily Corticosteroid Therapy
Brief Title: Safety Study of PI-0824 to Treat Pemphigus Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peptimmune (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: PI-001
Record Dates: First submitted 2003-07-03; First posted 2003-07-08 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-04

CONDITIONS: Pemphigus Vulgaris
MeSH Terms: conditions — Pemphigus

INTERVENTIONS:
Drug: PI-0824

SUMMARY:
The purpose of this study is to determine if the use of PI-0824 in patients with Pemphigus vulgaris is safe.

DETAILED DESCRIPTION:
Pemphigus vulgaris (PV) is an autoimmune disease affecting approximately 40,000 people worldwide. People with PV produce antibodies that attack the cells of the skin, resulting in blisters which, if left untreated, can lead to devastating infections and discomfort. Currently, most doctors who treat patients with PV will prescribe high-dose steroids and drugs that suppress the immune system in an effort to decrease the production of these antibodies. Unfortunately these medications are associated with serious and difficult side effects that often result in the discontinuation of their use. Peptimmune, Inc. has developed a new therapy for the treatment of PV, PI-0824. The goal of this therapy is to reduce the production of antibodies that cause PV blisters by acting only on the disease causing components of the immune system. It is hoped that use of PI-0824 will reduce or potentially eliminate the need for high dose steroids and drugs that suppress the immune system.

ELIGIBILITY:
Currently experiencing a stable disease course and medication regimen. Currently taking daily corticosteroid therapy for PV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2003-07; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California San Francisco, San Francisco, California
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - East Coast Clinical Research, Salisbury, Massachusetts
  - Stony Brook Dermatology Associates, East Setauket, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYU School of Medicine, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- See also: International Pemphigus Foundation — http://www.pemphigus.org